CLINICAL TRIAL: NCT02095301
Title: Herbal Extract Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: PEP-1320
Record Dates: First submitted 2014-03-10; First posted 2014-03-24 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Normal Controls

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Control plus herbal extract (Experimental): Control plus herbal extract
  Interventions: Other: Herbal Beverage
- Caffeine-free, carbonated soft drink (Placebo Comparator): Caffeine-free, carbonated soft drink

INTERVENTIONS:
Other: Herbal Beverage
  Arms: Control plus herbal extract

SUMMARY:
The objective of this study is to assess the effects of an herbal extract on mental energy in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 18-70 years of age, inclusive.
2. Subject has a body mass index (BMI) ≥17.0 and ≤32.9 kg/m2 at visit 1 (day -14 to -2).
3. Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history, and routine laboratory test results.
4. Subject is a non-smoker, defined as no tobacco use for ≥6 months prior to visit 1 (day -14 to -2).
5. Individual is willing to maintain a habitual diet and physical activity patterns throughout the study period.
6. Subject is willing to consume study product and standardized meals.
7. Individual is willing to abstain from caffeinated beverages and other caffeine-containing products for 12 h prior to all test visits (visits 2, 3, and 4; days 0, 3, and 6).
8. Subject is willing to abstain from alcohol consumption and avoid non-routine vigorous physical activity for 24 h prior to all test visits (visits 2, 3, and 4; days 0, 3, and 6).
9. Subject is willing to discontinue any vitamin/mineral or dietary supplements use for 2 weeks prior to visit 2 (day 0) and throughout the study period.
10. Subject is a female who is willing to schedule the randomization visit (visit 2, day 0) during the luteal phase of her menstrual cycle, defined as days 15 to the end of the cycle, where day 1 is the first day of menses, where appropriate.
11. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subject is unable to understand and/or perform required tests and questionnaires (i.e., subjects cannot complete the practice tests, or tasks).
2. Subject is color blind.
3. Subject has an abnormal laboratory test result of clinical significance, including, but not limited to creatinine ≥1.5 mg/dL and ALT or AST ≥1.5X upper limit of normal at visit 1 (day -14 to -2).
4. Subject has a known allergy or sensitivity to study products or any ingredients of the study products, standardized meals/snacks provided.
5. Subject has a gastrointestinal condition that could potentially interfere with absorption of the study product (e.g., inflammatory bowel syndrome, celiac disease, history of gastric bypass surgery).
6. Subject has diagnosed depression, schizophrenia, or dementia in the last 2 years prior to visit 1 (day -14 to -2).
7. Subject has a history or presence of clinically important cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, and/or stroke), renal, hepatic, endocrine (including type 1 or type 2 diabetes mellitus), pulmonary, biliary, pancreatic, or neurologic disorders.
8. Subject has extreme dietary habits (e.g., vegan, Atkins diet, very high protein).
9. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg as defined by the blood pressure measured at visit 1, (day -14 to -2). One re-test will be allowed on a separate day prior to visit 2 (day 0) for subjects whose blood pressure exceeds either of these cut points at visit 1.
10. Subject has a history or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
11. Subject has signs/symptoms of an active infection of clinical relevance (e.g., urinary tract or respiratory infection). Test visits (visits 2, 3, and 4; days 0, 3, and 6) will be re-scheduled to allow subject to be symptom-free of any type of systemic infection for at least 5 d.
12. Subject has recently used antibiotics (within 5 d of any test visit; Appendix 1). Test days (visits 2, 3, and 4; days 0, 3, and 6) will be rescheduled to allow the subject to be free of antibiotic therapy for at least 5 d.
13. Subject has a history of use of psychotropic medications within 6 months of visit 2 (day 0) and throughout study period.
14. Subject has used any other prescription medications, including over-the-counter medications within 2 weeks of visit 2 (day 0; Appendix 1) and throughout study period.
15. Subject has used any over-the-counter or prescription sleep aid products (including dietary supplements) within 2 weeks of visit 2 (day 0) and throughout study period.
16. Subject has a diagnosed sleep disorder (e.g., sleep apnea) or occupation where sleep during the overnight hours is irregular (e.g., 3rd shift or overnight workers).
17. Subject consumes excessive amounts of caffeine (>4 cups of caffeinated coffee/d or >400 mg caffeine/d from caffeine-containing products).
18. Subject is a female, who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source document.
19. Subject has a recent history of (within 12 months of screening; visit 1, day -14 to -2) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
20. Subject has been exposed to any non-registered drug product within 30 d prior to screening.
21. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Changes in the ratings from computer administered tasks within the domains of mood, short-term recognition memory, and attention from pre- to post-study product consumption and between treatment conditions of an herbal extract | 0-2 hours

SECONDARY OUTCOMES:
Measure plasma nutrient metabolites | 0-7 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Anil Samsong, Addison, Illinois, United States